CLINICAL TRIAL: NCT06467942
Title: Effects of Estrogen-like Chinese Medicine and Vaginal Lactobacillus on HPV Clearance and Vaginal Microbiota Change in Women With Persistent HPV Infection
Brief Title: Effects of Chinese Medicine and Lactobacillus in Persistent HPV Infection
Acronym: ELIMVLHPV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Mingzhu Li, Principal Investigator, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELIM-HPV2023
Record Dates: First submitted 2023-02-17; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Human Papilloma Virus Infection
MeSH Terms: conditions — Papillomavirus Infections | interventions — Lacteol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- observation group (No Intervention): Observation and follow-up only, no medication
- combined drug group (Experimental): Chinese medicine 5 days + Lactobacillus 5 days
  Interventions: Drug: Chinese medicine and Lactobacillus
- Single Chinese medicine group (Active Comparator): Chinese medicine group 10 days
  Interventions: Drug: Chinese medicine
- Single Lactobacillus group (Active Comparator): Lactobacillus group: 10 days
  Interventions: Drug: Lactobacillus

INTERVENTIONS:
Drug: Chinese medicine and Lactobacillus — combined drug group
  Other Names: Baofukang and Dingjunsheng
  Arms: combined drug group
Drug: Chinese medicine — Single Chinese medicine group
  Other Names: Baofukang
  Arms: Single Chinese medicine group
Drug: Lactobacillus — Single Lactobacillus group
  Other Names: Dingjunsheng
  Arms: Single Lactobacillus group

SUMMARY:
High risk human papillomavirus (hr-HPV) persistent infection is a high risk factor for cervical cancer. 85% to 90% of hr-HPV infections have the ability to clear on their own, while 10% to 15% of HPV persists further will lead to the development of high-grade intraepithelial lesions (HSIL) and even to invasive cervical cancer. Long-term follow-up results for persistent hr-HPV infection showed that cervical HSIL mostly occurred after 5-7 years of persistent hr-HPV infection, among which the risk of HPV16 and 18 was the highest, followed by HPV31 and 33. The role of the vaginal microbiome (CVM) in persistent hr-HPV infection has been increasingly valued, and women with persistent HPV infection that progresses to HSIL have a more unstable vaginal microenvironment. The previous study found that Lactobacillus vaginalis may contribute to HPV clearance by improving the vaginal microenvironment. In addition, previous studies have found that estrogen-like Chinese medicine could increase glycogen, improve mucosal estrogen levels, increase lactobacillus content, and promote HPV clearance. It is a challenge to make clinical management on when and how to intervene among hr-HPV persistent infection but whose pathology does not suggest HSIL. This study intends to analyze the correlation between the duration of HPV infection and the current vaginal microbiome, HPV load and PAX1 methylation in people with persistent HPV infection at different ages, and observe the changes of the above indicators after the administration of drugs to improve the vaginal microenvironment, which is helpful for preventing HPV persistent infection and developing into true precancerous lesions. It has the clinical and practical value of "preparing for a rainy day".

DETAILED DESCRIPTION:
1. Correlation of Previous Persistent HPV Infection Duration with Current CST, HPV Load, and PAX1 Methylation Participants: Select 240 women aged 25 and above who have had persistent high-risk HPV infection of the same type for 1 year or more but whose pathology does not indicate HSIL.

   Data Recording: Record the time of first confirmed HPV infection based on test reports.

   Initial Testing: After meeting the inclusion criteria, conduct initial tests for vaginal microbiota types (CST), HPV load, and PAX1 methylation.

   Correlation Analysis: Analyze the correlations based on different ages, menopausal status, and duration of HPV infection.
2. Changes in CST, HPV Load, and PAX1 Methylation After Treatment to Improve Vaginal Microenvironment

Study Design: Conduct a double-blind randomized medication trial with the participants divided into four groups:

Traditional Chinese Medicine Group: 10 days Lactobacillus Group: 10 days Combination Group: Traditional Chinese Medicine for 5 days + Lactobacillus for 5 days Control Group: Observation only, no medication Pre-Treatment: If applicable, treat any existing vaginitis before assigning medications.

Medication Regimen: Administer 10 consecutive days of vaginal medication each month, pausing during menstruation and resuming post-menstruation to complete the 10-day course. Sexual intercourse is prohibited during the medication period.

Follow-Up Testing: Conduct CST, HPV load, and PAX1 methylation tests at 6 and 12 months post-treatment.

Progression Monitoring: If HPV remains positive upon retesting, perform a colposcopy. Terminate the study and provide appropriate treatment if pathology progresses to HSIL.

ELIGIBILITY:
Inclusion Criteria:

* Women over 25 years of age with the same type of high-risk HPV infection lasting for more than 1 year, atypical squamous cell (ASCUS) or Low-grade squamous intraepithelial disease (LSIL) cytologically negative or undiagnosable, and pathological biopsy results negative or LSIL
* Consent to use the device for contraception during the study period;
* agree with medicine and follow-up management procedure.

Exclusion Criteria:

* High cytological risk, including atypical squamous cells (ASC-H),HSIL and atypical glandular cell (AGC), which could not rule out high-grade squamous intraepithelial lesions;
* pathological biopsy for HSIL and above;
* for any drug allergies;
* pregnancy or lactation

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — physical examination was female
Enrollment: 240 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
community state type (CST) | Change of CST at 6 months and 12 months after medication
  Vaginal microflora type
HPV VL | Change of HPV VL at 6 months and 12 months after medication
  HPV viral load
PAX1 methylation test | Change of PAX1 methylation test at 6 months and 12 months after medication
  Pairing box gene1 methylation test

SECONDARY OUTCOMES:
Complete remission (CR) | Change of CR at 6 months and 12 months after medication
  HPV subtypes with persistent infection turned negative at 6 and 12 months or positive at 6 months, and negative at 12 months
Partial remission (PR) | Change of PR at 6 months and 12 months after medication
  Partial response (PR) : HPV subtypes with persistent infection turned negative at 6 months and returned positive at 12 months
No response (NR) | Change of NR at 6 months and 12 months after medication
  HPV subtypes with persistent infection were positive at both follow-up visits

CONTACTS AND LOCATIONS:
Overall Officials: Mingzhu Li, Principal Investigator — Peking University People's Hosptial
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China